CLINICAL TRIAL: NCT01537120
Title: Evaluation of Continuous Glucose Monitoring as a Tool to Measure Glucoregulatory Effects of a Twice Daily Oral Insulin Secretagogue
Brief Title: Evaluation of Continuous Glucose Monitoring in Participants With Type 2 Diabetes Mellitus (MK-0000-258 AM2)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 0000-258
Record Dates: First submitted 2011-12-22; First posted 2012-02-23 (Estimated); Results first posted 2013-12-03 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

STUDY DESIGN:
Who Masked: Participant

ARMS (1):
- Placebo → Vildagliptin (Experimental): Participants received placebo tablets orally, twice a day for 3 weeks, and then over the next 12 weeks received vildagliptin 50 mg tablets orally, twice daily
  Interventions: Drug: Vildagliptin; Drug: Placebo

INTERVENTIONS:
Drug: Vildagliptin
Drug: Placebo

SUMMARY:
This trial will attempt to develop the use of Continuous Glucose Monitoring (CGM) as a tool for the evaluation of both new and existing pharmacological treatments for type 2 diabetes, using the twice daily administered dipeptidyl peptidase-4 (DPP4) inhibitor, vildagliptin as a probe. The primary hypothesis is that two weeks of treatment with 50 mg of oral Vildagliptin, twice daily will lead to a statistically significant decrease in 24 hour weighted-mean glucose (WMG) relative to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 2 diabetes mellitus on a clinical regimen that is metformin alone, up to a maximum of 3 gram per day, on a background of lifestyle measures, and has a Hemoglobin A1C at screening of > 7%.
* If on antihyperglycemic therapy with both metformin and sulfonylurea with a Screening Visit/Visit 1 Hemoglobin A1C of >= 6.5% and =< 7.5%, should then discontinue sulfonylurea usage and undergo washout of sulfonylurea.

Exclusion Criteria:

* History of either stroke, chronic seizures or major neurological disorder within the last 6 months.
* Untreated hypertension with a blood pressure of > 160/95 mmHg.
* History of neoplastic disease within the past 5 years.
* History of hypersensitivity to vildagliptin or other DPP4 inhibitors.
* Had major surgery, or donated or lost 1 unit (500 mL) of blood, or participated in another investigational study within 4 weeks prior to screen.
* Used any illicit drug or abusively used alcohol within the past 3 months.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-12; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After enrollment, participants previously treated with both metformin and sulfonylurea, discontinued sulfonylurea usage and underwent washout of sulfonylurea over a period of 8 weeks prior to treatment. Non-washout participants were enrolled on a clinical regimen of metformin alone.
Period: Enrolled
Arm/Group | Placebo → Vildagliptin
Started | 25
Completed | 25
Not Completed | 0
Period: 8 Weeks Washout
Arm/Group | Placebo → Vildagliptin
Started | 25
Completed | 24
Not Completed | 1
Not completed — Inclusion/exclusion criteria not met | 1
Period: 3 Weeks Placebo
Arm/Group | Placebo → Vildagliptin
Started | 24
Completed | 23
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: 12 Weeks Vildagliptin
Arm/Group | Placebo → Vildagliptin
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Placebo → Vildagliptin
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 24

OUTCOME MEASURES:

1. Primary Outcome: 24 Hour Weighted Mean Glucose (WMG) At 2 Weeks
Description: The 24 hour WMG was measured after 2 weeks of placebo treatment, and again after 2 weeks of vildagliptin treatment. Glucose was measured over a 24 hour period by having participants wear two continuous glucose monitors (CGM), which produced an average glucose value approximately every 5 minutes. Using these values, the concentration of glucose was calculated from Area Under the Curve 0-24 hours (AUC 0-24hr), and was expressed as 24 hour WMG.
Time Frame: At 2 weeks after Placebo treatment and again at 2 weeks after Vildagliptin treatment
Population: Per-Protocol Population: all participants who complied with the assigned medication during each period of study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/dL
Groups:
- Placebo: Placebo tablets twice daily for 3 weeks
- Vildagliptin: Vildagliptin tablets 50 mg twice daily for 12 weeks
Arm/Group | Placebo | Vildagliptin
Number analyzed (Participants) | 24 | 23
mg/dL | 126.9 (16) | 114.2 (17)
Statistical Analysis 1: Comparison: Placebo vs Vildagliptin; Test type: Superiority or Other; Geometric Mean Ratio = 0.91, 90% CI 2-sided [0.85 to 0.96]

2. Secondary Outcome: Hemoglobin A1C (HbA1C) At 2 Weeks
Description: Blood samples were taken after 2 weeks of placebo treatment, and again after 2 weeks of vildagliptin treatment to measure the percentage of glycated hemoglobin, HbA1C. Units are therefore presented as HbA1c (%).
Time Frame: At 2 weeks after Placebo treatment and again at 2 weeks after Vildagliptin treatment
Population: Per-Protocol Population: all participants who complied with the assigned medication during each period of study.
Measure: Mean (Standard Deviation); unit: HbA1c (%)
Arm/Group | Placebo | Vildagliptin
Number analyzed (Participants) | 24 | 23
HbA1c (%) | 7.12 (0.54) | 6.82 (0.55)
Statistical Analysis 1: Comparison: Placebo vs Vildagliptin; Test type: Superiority or Other; Least Squares Mean Difference = -0.30, 90% CI 2-sided [-0.36 to -0.23]

3. Secondary Outcome: HbA1C At 12 Weeks
Description: Blood samples were taken after 2 weeks of placebo treatment, and again after 12 weeks of vildagliptin treatment to measure the percentage of glycated hemoglobin, HbA1C. Units are therefore presented as HbA1c (%).
Time Frame: At 2 weeks after Placebo treatment and again at 12 weeks after Vildagliptin treatment
Population: Per-Protocol Population: all participants who complied with the assigned medication during each period of study.
Measure: Mean (Standard Deviation); unit: HbA1c (%)
Arm/Group | Placebo | Vildagliptin
Number analyzed (Participants) | 24 | 23
HbA1c (%) | 7.12 (0.54) | 6.66 (0.74)
Statistical Analysis 1: Comparison: Placebo vs Vildagliptin; Test type: Superiority or Other; Least Squares Mean Difference = -0.46, 90% CI 2-sided [-0.62 to -0.30]

ADVERSE EVENTS:
Groups:
- Vildagliptin 50 mg: Vildagliptin tablets 50 mg twice daily for 12 weeks
Arm/Group | Vildagliptin 50 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 8/23 | 6/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vildagliptin 50 mg (N=23) | Placebo (N=24)
Reaction CGM Site (General disorders) | 2 (2) | 2 (2)
Reaction site cannula (General disorders) | 3 (4) | 5 (5)
Tiredness (General disorders) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 4 (4)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 4 (4) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission.